CLINICAL TRIAL: NCT05902988
Title: A Phase I/II Study of VLS-1488 (an Oral KIF18A Inhibitor) in Subjects With Advanced Cancer
Brief Title: A Phase I/II Study of VLS-1488 in Subjects With Advanced Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Volastra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VLS-1488-2201
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; High Grade Serous Adenocarcinoma of Ovary; Squamous Non-small-cell Lung Cancer; Triple Negative Breast Cancer; Head and Neck Squamous Cell Carcinoma; Ovarian Carcinosarcoma; Uterine Carcinosarcoma; Uterine Serous Carcinoma; Endometrium Cancer; Chromosomal Instability
Keywords: KIF18A Inhibitor; HGSOC; TNBC; HNSCC; sqNSCLC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Endometrial Neoplasms; Chromosomal Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: Dose Escalation Cohorts (Experimental): Subjects will be enrolled at various doses and/or schedules of VLS-1488. These Dose Escalation Cohorts will be utilized to identify the MTD and to select dose levels for Dose Expansion.
  Interventions: Drug: VLS-1488
- Dose Escalation: Backfill Cohorts (Experimental): Additional subjects may be enrolled at any dose level that does not meet de-escalation or elimination rules per the BOIN design. These Backfill Cohorts will be utilized to build additional data to support selection of doses and/or tumor types for further study in Dose Expansion.
  Interventions: Drug: VLS-1488
- Dose Expansion: Exploration Cohorts (Experimental): Subjects with a selected single tumor type will be randomized 1:1 into Exploration Cohorts at two or more dose levels of interest. A subset of subjects will have additional assessments to examine the potential for VLS-1488 to interact with other drugs and the effect of food on VLS-1488 absorption.
  Interventions: Drug: VLS-1488
- Dose Expansion: Development Cohorts (Experimental): Subjects with other tumor types will be enrolled at a single dose level of interest. These Development Cohorts will be utilized to examine the preliminary efficacy of VLS-1488 in various tumor types.
  Interventions: Drug: VLS-1488

INTERVENTIONS:
Drug: VLS-1488 — VLS-1488 tablets will be given orally.

SUMMARY:
This is a first-in-human phase I/II study to examine the safety, tolerability and preliminary efficacy of VLS-1488 in subjects with advanced cancers.

DETAILED DESCRIPTION:
This a first-in-human phase I/II study designed to assess the safety, tolerability and preliminary efficacy of VLS-1488 monotherapy and consists of two parts: Dose Escalation and Dose Expansion.

Dose Escalation will examine the safety and tolerability of VLS-1488 in different solid tumor types at various dose levels through a series of Dose Escalation and Backfill Cohorts to identify the Maximum Tolerated Dose (MTD) and to select dose levels for Dose Expansion. The criteria for dose (de-)escalation will be based on a Bayesian Optimal Interval (BOIN) design.

Dose Expansion will examine the safety, tolerability, Drug Drug Interaction (DDI) risk, Food Effect (FE) and preliminary efficacy of VLS-1488 in different tumor types and/or dose levels of interest through various expansion cohorts.

VLS-1488 will be given orally in 28-day cycles. Dosing will be continued until disease progression, unacceptable toxicity, withdrawal of consent, or other stopping criteria are met.

ELIGIBILITY:
Key Inclusion Criteria:

* All Parts: Age ≥ 18 years, ECOG Performance Status ≤ 1, at least 1 site of measurable disease evaluable by CT scan or MRI per RECIST 1.1, able to take oral medication without alteration
* Dose Escalation: No available therapeutic options to provide clinically meaningful benefits in the following tumor types: High Grade Serous Ovarian Cancer, Squamous Non -Small Cell Lung Cancer, Triple Negative Breast Cancer, Gastric Adenocarcinoma (not EBV+), Colorectal, Esophageal Squamous Cell Carcinoma, Esophageal Adenocarcinoma, Gastroesophageal Junction, Bladder (transitional cell), Head and Neck Squamous Cell Carcinomas (not nasopharynx, sinonasal or lip), Ovarian Carcinosarcoma, CN-high Endometrial/Uterine
* Dose Expansion: Must have been previously treated with several lines of standard of care treatment specified in the protocol in the following tumor types: High Grade Serous Ovarian Cancer, Squamous Non-Small Cell Lung Cancer, Triple Negative Breast Cancer, Gastric Adenocarcinoma (not EBV+), Colorectal, Esophageal Squamous Cell Carcinoma, Esophageal Adenocarcinoma, Head and Neck Squamous Cell Carcinomas (not nasopharynx, sinonasal or lip), CN-high Endometrial/Uterine

Key Exclusion Criteria:

* MSI-H, dMMR, POLE gene hotspot mutated, or known hypermutator phenotype
* Previously received KIF18A inhibitor
* Current CNS metastases or leptomeningeal disease
* Cardiac parameters: MI or stroke ≤ 1 year, unstable angina/PE/DVT/CABG ≤ 6 months, NYHA Class ≥ II, LVEF < 50%
* Inability to comply with concomitant medication restrictions with respect to strong inhibitors and inducers of CYP3A, and clinical inhibitors of MDR1 (P-gp) and BCRP
* Any clinically significant ascites or pleural effusions at time of enrollment, or any therapeutic paracentesis or thoracentesis within 28 days of planned first dose of study drug
* Bowel obstruction or GI perforation within 6 months of planned first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of Dose Limiting Toxicities (DLTs) in DLT-evaluable subjects | Up to 12 months
Dose Escalation: Determination of the MTD of VLS-1488 | Up to 12 months
Dose Escalation: Frequency of Serious Adverse Events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | Up to 12 months
Dose Escalation: Frequency of Treatment-related Adverse Events (AEs) graded per NCI-CTCAE version 5.0 | Up to 12 months
Dose Escalation: Frequency of Treatment-Emergent AEs (TEAEs) graded per NCI-CTCAE version 5.0 | Up to 12 months
Dose Escalation: Frequency of Dose Interruptions and Permanent Treatment Discontinuations | Up to 12 months
Dose Expansion: Frequency of Trigger Events (TEs) | Up to 18 months
Dose Expansion: Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 18 months

SECONDARY OUTCOMES:
Dose Escalation: ORR as assessed by RECIST version 1.1 | Up to 12 months
Dose Expansion: Frequency of SAEs graded according to NCI-CTCAE version 5.0 | Up to 18 months
Dose Expansion: Frequency of Treatment-related AEs graded according to NCI-CTCAE version 5.0 | Up to 18 months
Dose Expansion: Frequency of TEAEs graded according to NCI-CTCAE version 5.0 | Up to 18 months
Dose Expansion: Frequency of Dose Interruptions and Permanent Treatment Discontinuations | Up to 18 months
Dose Expansion: Area Under the Plasma Concentration-Time Curve (AUC) of Midazolam and its metabolite 1'-hydroxymidazolam | Up to 18 months
Dose Expansion: Maximum Plasma Concentration (Cmax) of Midazolam and its metabolite 1'-hydroxymidazolam | Up to 18 months
Dose Expansion: Evaluation of CA-125 response by Gynecologic Cancer InterGroup (GCIG) criteria (High Grade Serous Ovarian Cancer only) | Up to 18 months
Dose Escalation & Dose Expansion: Duration of Response (DOR) as assessed by RECIST version 1.1 | Up to 32 months
Dose Escalation & Dose Expansion: Disease Control Rate (DCR) as assessed by RECIST version 1.1 | Up to 32 months
Dose Escalation & Dose Expansion: Progression Free Survival (PFS) as assessed by RECIST version 1.1 | Up to 32 months
Dose Escalation & Dose Expansion: Cmax of VLS-1488 | Up to 32 months
Dose Escalation & Dose Expansion: AUC of VLS-1488 | Up to 32 months
Dose Escalation & Dose Expansion: Trough Concentration (Ctrough) of VLS-1488 | Up to 32 months
Dose Escalation & Dose Expansion: Time to Maximum Plasma Concentration (Tmax) of VLS-1488 | Up to 32 months
Dose Escalation & Dose Expansion: Ratio of Total Cholesterol to 4β-hydroxycholesterol in plasma | Up to 32 months
Dose Escalation & Dose Expansion: Increase in the number of Phospho-Histone 3 positive tumor cells | Up to 32 months
Dose Escalation & Dose Expansion: Frequency of Micronucleated Reticulocytes in blood | Up to 32 months
Dose Escalation & Dose Expansion: Increase in Micronuclei in Circulating Tumor Cells | Up to 32 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Kellogg Cancer Center, Evanston, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Women & Infants Hospital, Providence, Rhode Island
  - M.D. Anderson Cancer Center, Houston, Texas
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided